CLINICAL TRIAL: NCT05297461
Title: Impact of Community Pharmacists' Medication Review on Medication Use Related Problems Among Older Adults in Penang: A Pilot Randomised Controlled Study
Brief Title: Impact of Medication Review by Community Pharmacists
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Monash University Malaysia (Other)
Responsible Party: Principal Investigator, Christina Christopher, Principal Investigator, Monash University Malaysia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: MedRev
Record Dates: First submitted 2022-03-17; First posted 2022-03-28 (Actual); Last update posted 2023-10-31 (Actual); Status verified 2023-10

CONDITIONS: Aging
MeSH Terms: interventions — Medication Review

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Medication Review (Experimental): The intervention group will receive medication review intervention which includes reviewing older adults' medications and identifying any drug-related problems.
  Interventions: Other: Medication review
- Standard Care (No Intervention): The standard care includes the current existing care provided to patients in the community pharmacy.

INTERVENTIONS:
Other: Medication review — Community pharmacy benchmarking guideline Pharmaceutical Services Division provides guidelines for medication review in community pharmacy settings in Malaysia
  Arms: Medication Review

SUMMARY:
The aging population size has been enlarging globally. A higher number of older adults means a higher number of medication use. It is estimated that older adults are the largest medication consumers.That would result in various medication use problems which provide a link between polypharmacy, inappropriate medication, and deprescribing.[2] Primary health care providers especially community pharmacists are often the first point of healthcare towards older adults.[3] Various interventions are being carried out by community pharmacies to determine an optimal outcome on medication usage.

Medication review intervention is a clinical process where a pharmacist reviews a patient's medication, identifies any drug-related problems and suggests strategies to reduce the medication use problems. Medication review is being utilized in various countries especially in Organisation for Economic Co-operation and Development (OECD )regions ie Australia, New Zealand, the United Kingdom, and the United States of America, and the pharmacist were remunerated for the service. Although medication review is widely searched intervention globally, the scope for intervention is lacking in low and middle-income countries.

Community pharmacy is regarded as the first point of care of primary health care in a community for older adults. A systemic review search on community pharmacist-led intervention among the aging population has demonstrated medication adherence improvement outcomes. Consequently, community pharmacists can reduce medication use problems in different settings in the community in various ways and contribute to the patients' overall well-being and health-related quality of life.

There is a lack of information in Malaysia due to the fragmented health care system where there is no continuity of care between the public and private sectors. During this pandemic outbreak, when most countries suffer critical health care points, much effort and pharmaceutical care should be delivered towards older adults to reduce the current burden. This study assesses the feasibility of medication review for older adults at the community pharmacy level and identifies any medication-related problems in Penang state. The significance of this study is improving medication use among older adults at a primary care level and will probably upgrade the quality of the Malaysian health care system by providing some program and policy level solutions towards the problems.

DETAILED DESCRIPTION:
* Before the initiation of the study, the community pharmacy involved or volunteered from intervention groups in Penang, Malaysia will undergo half-day training on a structured medication review plan and the study process.
* Control groups pharmacies will undergo a briefing of the study process only.
* A validated survey MedUseQ questionnaire will be administered to each respondent from both intervention and control groups prior to the intervention.
* Medication review intervention will then be performed only for the intervention group.
* A pharmacist will review the medications of those in the intervention group and tried to resolve any drug-related problems encountered by the participants. In addition, the pharmacist will conduct a question-answer session with the participants to enhance older adults' knowledge and awareness of their medications.
* Immediate post-intervention knowledge questions related to their medications name and dose, timing and interval of dose, medication indication, and possible side effects.
* Intervention groups will be followed up at two months and four months through a phone call or face to face. Follow-up will include detecting any medication-related problems among participants, updating their current medication regime, and to further clarifying any query from them.
* Meanwhile, the control group will not be going under follow-up. Only the number of drug related problems will be recorded
* All participants will then be followed six months of post-intervention and will be given again the MedUseQ survey to compare the difference between baseline and post-intervention.
* Data collection will be conducted at baseline and six months after the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Patients above 60 years old Patients who have chronic disease ie diabetes, hypertension, cardiovascular
* Patients who have been patronizing the pharmacy for the purchase of at least one prescription medication for the past three months.
* Patients be able to converse, read and understand the Malay language or English language.
* Access to a telephone or mobile phone or internet
* The patients must understand the study process, agree to participate in this study, and sign the informed consent

Exclusion Criteria:

* Patient who are unable to converse, read and understand Malay or English language
* Patients who unable to give their consent

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2022-06-30 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2023-01-30 (Actual)

PRIMARY OUTCOMES:
Assessing feasibility: intervention time | 6 months
  Length of intervention (minutes)
Assessing feasibility: Number of staffs | 6 months
  Number of staffs
Assessing feasibility: Access to prescribers | 6 months
  Number of prescribers contacted
Type and number medication-related problem | 6 months
  1. Number of inappropriate medications (Based on Beer's criteria)
  2. Number of medications
  3. Adverse drug reactions detected
  4. Drug-drug interaction
  5. Improper medication administration
  6. Incorrect dose and frequency of medications

CONTACTS AND LOCATIONS:
Locations (1):
- Northern MCPG, George Town, Pulau Pinang, Malaysia

REFERENCES:
- [Background] Marek KD, Antle L. Medication Management of the Community-Dwelling Older Adult. In: Hughes RG, editor. Patient Safety and Quality: An Evidence-Based Handbook for Nurses. Rockville (MD): Agency for Healthcare Research and Quality (US); 2008 Apr. Chapter 18. Available from http://www.ncbi.nlm.nih.gov/books/NBK2670/ PMID 21328769
- [Background] Mangin D, Garfinkel D. Foreword to the first special collection: Addressing the invisible iatrogenic epidemic: the role of deprescribing in polypharmacy and inappropriate medication use. Ther Adv Drug Saf. 2019 Oct 21;10:2042098619883156. doi: 10.1177/2042098619883156. eCollection 2019. No abstract available. PMID 31673327
- [Background] Ramli A, Taher S. Managing chronic diseases in the malaysian primary health care - a need for change. Malays Fam Physician. 2008 Apr 30;3(1):7-13. eCollection 2008. PMID 25606105
- [Background] Blenkinsopp A, Bond C, Raynor DK. Medication reviews. Br J Clin Pharmacol. 2012 Oct;74(4):573-80. doi: 10.1111/j.1365-2125.2012.04331.x. PMID 22607195
- [Background] Lee E, Braund R, Tordoff J. Examining the first year of Medicines Use Review services provided by pharmacists in New Zealand: 2008. N Z Med J. 2009 Apr 24;122(1293):3566. PMID 19448788
- [Background] Ramalho de Oliveira D, Brummel AR, Miller DB. Medication therapy management: 10 years of experience in a large integrated health care system. J Manag Care Pharm. 2010 Apr;16(3):185-95. doi: 10.18553/jmcp.2010.16.3.185. PMID 20331323
- [Background] Benrimoj SI, Roberts AS. Providing patient care in community pharmacies in Australia. Ann Pharmacother. 2005 Nov;39(11):1911-7. doi: 10.1345/aph.1G165. Epub 2005 Oct 11. PMID 16219897
- [Background] Beuscart JB, Petit S, Gautier S, Wierre P, Balcaen T, Lefebvre JM, Kambia N, Bertoux E, Mascaut D, Barthelemy C, Cuny D, Puisieux F, Decaudin B. Polypharmacy in older patients: identifying the need for support by a community pharmacist. BMC Geriatr. 2019 Oct 21;19(1):277. doi: 10.1186/s12877-019-1276-y. PMID 31638909
- [Derived] Christopher CM, Blebil AQ, Bhuvan KC, Alex D, Ibrahim MIM, Ismail N, Cheong MWL. Assessing feasibility of conducting medication review with follow-up among older adults at community pharmacy: a pilot randomised controlled trial. Int J Clin Pharm. 2024 Aug;46(4):843-853. doi: 10.1007/s11096-024-01711-3. Epub 2024 Apr 18. PMID 38635115